CLINICAL TRIAL: NCT02829125
Title: Influence of Postoperative Rehabilitation and Pre- and Postoperative Physical Activity in Abdominal Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6254
Record Dates: First submitted 2016-06-17; First posted 2016-07-12 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2015-01

CONDITIONS: Abdominal Injuries
Keywords: Early rehabilitation; abdominal surgery; ERAS
MeSH Terms: conditions — Abdominal Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The concept of early rehabilitation (ERAS: enhanced after-surgery recovery) was introduced by Kehlet et al. in 1995, as part of the colon surgery. This program is a support for patients combining laparoscopic surgery, epidural analgesia, early refeeding and rapid mobilization of patients. This strategy targets multiple elements (20 items) to support pre-, intra- and postoperative patients. This reduces the pain and the different organ dysfunction induced by surgical stress significantly decreasing length of hospital stay, postoperative morbidity and costs.

Furthermore, early mobilization of patients is fundamental to the ERAS method. Few studies have analyzed the influence of preoperative exercise on postoperative rehabilitation.

ELIGIBILITY:
Inclusion criteria

1. non-cancerous and cancerous pathology
2. signed Consent
3. Every patient operated on a scheduled or emergency abdominal surgery

Exclusion criteria

1. inability to give informed about information
2. minor Patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing abdominal surgery
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-01-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
quality of life questionnaire | before and after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe STEINMETZ, MD, Study Director — University Hospital, Strasbourg, France; Benoît ROMAIN, MD, PhD, Principal Investigator — University Hospital, Strasbourg, France; Serge ROHR, MD, PHD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Service de Chirurgie Digestive - Hôpital de Hautepierre, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No